CLINICAL TRIAL: NCT00802841
Title: A Randomized Phase Lll Study of Imatinib Dose Optimization Compared With Nilotinib in Patients With Chronic Myelogenous Leukemia and Suboptimal Response to Standard-dose Imatinib
Brief Title: Randomized Phase Lll Study of Imatinib Dose Optimization vs Nilotinib in CML Patients With Suboptimal Response to Imatinib
Acronym: LASOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2404; 2008-007054-35 (EudraCT Number)
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic; Myelogenous; Leukemia; CML; Chronic Phase; Suboptimal Response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Bronchiolitis Obliterans Syndrome; Leukemia | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (Experimental): Participants received 400 mg nilotinib twice daily (BID).
  Interventions: Drug: nilotinib
- Imatinib (Active Comparator): Participants received 600 mg imatinib once daily (QD).
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: nilotinib — Supplied as 200 mg tablets
  Other Names: Tasigna
  Arms: Nilotinib
Drug: imatinib — Supplied as 100 mg and 400 mg tablets
  Other Names: Gleevec/Glivec
  Arms: Imatinib

SUMMARY:
There is no available data on the clinical benefit of dose escalation for patients with suboptimal response to imatinib, and patients may still improve their response with continuation of therapy at the standard dose as shown in the IRIS trial after 5 years of follow-up. However, there is no data yet regarding the potential benefit of using nilotinib in the group of patients with suboptimal response. In this study, the efficacy of nilotinib 400mg BID will be compared to imatinib 600mg QD.

DETAILED DESCRIPTION:
The comparative efficacy between imatinib dose escalation (600 mg QD) and nilotinib (400 mg BID), in terms of CCyR after 6 months, for patients with CML in chronic phase with suboptimal response to imatinib standard dose will be determined.

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥ 18 years old;
2. ECOG of 0, 1, or 2;
3. Ph+ CML in CP defined as:

   * <15% blasts in peripheral blood or bone marrow;
   * <30% blasts + promyelocytes in peripheral blood or bone marrow;
   * <20% basophils in the peripheral blood;

     •≥100x109/L (≥ 100,000/mm3) platelets;
   * no evidence of extramedullary leukemia involvement, with the exception of hepatosplenomegaly;
4. SoR to 400 mg imatinib, defined as (min of 20 metaphases):

   * No cytogenetic response at ≥ 3 to <6 months (> 95% Ph+ metaphases);or
   * No PCyR at ≥ 6 to <12 months (36 to 95% Ph+ metaphases on bone marrow); or
   * No CCyR at ≥ 12 to <18 months (1 to 35% Ph+ metaphases on bone marrow); Confirmation of SoR by FISH is allowed if BMK is done outside the screening window up to 4 wks.
5. 400mg/daily imatinib (no higher doses) for at least 3months but no longer than 18 months;
6. Previous use of IFN, taken prior to imatinib treatment, is allowed at a maximum of 90 days unless reason for switch from IFN to imatinib was intolerance.
7. Parameters must be present:

   * Creatinine <2.0 X ULN
   * Total bilirubin <1.5 X ULN (< 3.0 X ULN if related to disease);
   * SGOT and SGPT < 2.5 X ULN;
   * Serum lipase ≤1.5 X ULN;
   * Alkaline phosphatase ≤2.5 X ULN
   * Serum potassium, phosphorus, magnesium and calcium ≥ LLN or corrected to WNL with supplements prior to first dose of study drug;
8. Written informed consent prior to any study procedures being performed.

Exclusion criteria:

1. Prior accelerated phase including clonal evolution or blast crisis CML;
2. Prior therapy with imatinib in combination with any other CML drug other than Hydroxyurea and/or Anagrelide;

4.Imatinib therapy started more than 12 months after the date of the original diagnosis; 5.Unable to tolerate imatinib at 400mg; 6.Previous treatment with any other tyrosine kinase inhibitor except Glivec and/or CML therapy other than IFN, hydroxyurea, and /or anagrelide; 7.Myelotoxicity ≥ Grade 2 present at the time of randomization, 8.Previously documented T315I mutations; 9.Impaired cardiac function including one of these:

* Long QT syndrome or family history of long QT syndrome
* Clinically significant resting brachycardia (<50 bpm)
* QTcF >450 msec on screening ECG (using the QTcF formula). If QTc >450 and electrolytes are not with normal ranges, electrolytes should be corrected and then the patient rescreened for QTc to certify QTc <450 msec;
* Myocardial infarction ≤ 12 months prior to the first dose of study drug;
* Other clinically significant heart disease (e.g., CHF, uncontrolled hypertension, unstable angina, significant ventricular or atrial tachyarrhythmias) 10. Impairment of GI function or disease that may significantly alter the absorption of study drug; 11. Treated with strong CYP3A4 inhibitors that cannot be either discontinued or switched to a different medication prior to starting study drug; 12.Currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug; 13.History of previous acute pancreatitis within one year of study entry or medical history of chronic pancreatitis; 14.Known cytopathologically confirmed CNS 15.Women who are pregnant, breast feeding or of a childbearing potential without a negative urine pregnancy test at screening. Female patients of childbearing potential unwilling to use effective contraceptive precautions throughout the trial and for 3 months post trial end. Post-menopausal women must be ammenorrheic for at least 12 months to be considered of non-childbearing potential; 16. History of another primary malignancy that is currently clinically significant or currently requires active intervention; 17.Any other clinically significant medical or surgical condition which, according to investigators' discretion, should preclude participation; 18.Use of investigational agent within 28 days prior to enrollment; 19.Patients unwilling or unable to comply with the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2009-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- Argentina (3):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Rio Negro, Viedma
- Brazil (10):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Cuiaba, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Jaú, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- China (6):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Shanghai
- Colombia (2):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- India (7):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Mumbai 400 020
  - Novartis Investigative Site, New Delhi
- Mexico (3):
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Wroclaw
- Russia (8):
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Yekaterinburg
- Venezuela (2):
  - Novartis Investigative Site, Caracas, Distrito Federal
  - Novartis Investigative Site, Maracaibo, Zulia

REFERENCES:
- [Derived] Cortes JE, De Souza CA, Ayala M, Lopez JL, Bullorsky E, Shah S, Huang X, Babu KG, Abdulkadyrov K, de Oliveira JSR, Shen ZX, Sacha T, Bendit I, Liang Z, Owugah T, Szczudlo T, Khanna S, Fellague-Chebra R, le Coutre PD. Switching to nilotinib versus imatinib dose escalation in patients with chronic myeloid leukaemia in chronic phase with suboptimal response to imatinib (LASOR): a randomised, open-label trial. Lancet Haematol. 2016 Dec;3(12):e581-e591. doi: 10.1016/S2352-3026(16)30167-3. PMID 27890073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in 1:1 ratio to imatinib 600 mg QD or nilotinib 400 mg BID for a 2 year study period.
Pre-assignment Details: Cross-over from one arm to the other was allowed for intolerant patients anytime during treatment, patients who failed to achieve CCyR after 6 months of treatment, loss of response, loss of CHR, loss of best achieved cytogenetic response any time during treatment, or other reason approved by the Study Management Committee.
Groups:
- Imatinib: Participants receievd 600 mg imatinib once daily (QD).
Period: Overall Study
Arm/Group | Nilotinib | Imatinib
Started | 96 | 95
Full Analysis Set | 96 | 95
Safety Set | 96 | 93
Cross-over Set | 13 | 56
Completed | 0 | 0
Not Completed | 96 | 95
Not completed — Administrative problems | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 1 | 2
Not completed — Adverse Event | 8 | 2
Not completed — Disease progression | 7 | 3
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Protocol deviation | 2 | 6
Not completed — Treatment duration completed | 66 | 76

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib | Imatinib | Total
Number analyzed (Participants) | 96 | 95 | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (14.47) | 44.2 (15.02) | 44.4 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 37 | 79
  Male | 54 | 58 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR)
Description: CCyR was assessed from bone marrow samples. CCyr was defined as having 0% Philadelphia positive (Ph+) chromosome metaphases in bone marrow.
Time Frame: 6 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Percentage of participants | 50.0 | 42.1
Statistical Analysis 1: Comparison: Nilotinib vs Imatinib; Test type: Superiority or Other; p = 0.3106, Fisher Exact

2. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR)
Description: MMR was defined as having a fusion gene of the Bcr and Abl genes of (BCR-ACL) less than or equal to 0.1% on the International Scale (IS).
Time Frame: 12 and 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Percentage of participants
  12 months | 36.5 | 25.3
  24 months | 37.5 | 35.8

3. Secondary Outcome: Percentage of Participants With CCyr
Description: as for outcome 1
Time Frame: 12 and 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Percentage of participants
  12 months | 53.1 | 55.8
  24 months | 51.0 | 61.1

4. Secondary Outcome: Time to CCyR
Description: Time to CCyR was defined as time from date of randomization to date of first documented CCyR.
Time Frame: 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Months | 5.55 [5.52 to 5.98] | 5.85 [5.59 to 11.04]

5. Secondary Outcome: Duration of CCyR
Description: Duration of CCyR was defined as time from the date of ransomization to the date of first loss of CCyR or death, whichever came first.
Time Frame: 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Months | NA [NA to NA] — The median duration of CCyr was not achieved because there were not enough number of events. | 17.2 [17.2 to NA] — There were not enough events to calculate the upper limit of the 95% Confidence Interval (CI).

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of documented disease progression to accelerated phase or blast crisis (AP/BC), or death due to any cause.
Time Frame: 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Months | NA [NA to NA] — The median PFS time was not achieved. | NA [NA to NA] — The median PFS time was not achieved.

7. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from the date of randomization to the date of the first occurrence of any of the following: loss of Complete Hematological Response (CHR), loss of Partial Cytogenetic Response (PCyR), loss of CCyR, death on treatment or progression to AP/BC.
Time Frame: 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Months | NA [NA to NA] — The median EFS time was not achieved.. | 24.3 [23.8 to NA] — There were not enough events to calculate the upper limit of the 95% CI.

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from date of randomization to the date of the death.
Time Frame: 24 months
Population: Full Analysis Set: The FAS included all participants to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 96 | 95
Months | NA [NA to NA] — The median OS time was not achieved because there were not enough number of events. | 25.7 [NA to NA] — The median was estimated, but the standard error could not be estimated due to the limitation of the Kaplan Meier method where there were too few events and the last participant had a death. Therefore, the 95% CI could not be calculated.

ADVERSE EVENTS:
Groups:
- Cross-over to Nilotinib: Nilotinib 400 mg BID
- Cross-over to Imatinib: 600 mg QD
Arm/Group | Nilotinib | Imatinib | Cross-over to Nilotinib | Cross-over to Imatinib
Serious Adverse Events (participants affected / at risk) | 11/96 | 9/93 | 4/56 | 1/13
Other Adverse Events (participants affected / at risk) | 80/96 | 61/93 | 44/56 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=96) | Imatinib (N=93) | Cross-over to Nilotinib (N=56) | Cross-over to Imatinib (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Malaria antibody test positive (Investigations) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=96) | Imatinib (N=93) | Cross-over to Nilotinib (N=56) | Cross-over to Imatinib (N=13)
Anaemia (Blood and lymphatic system disorders) | 11 | 18 | 10 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 10 | 22 | 9 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 6 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 23 | 13 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 24 | 13 | 3
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 10 | 0 | 0
Papilloedema (Eye disorders) | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 2 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 15 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 14 | 4 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 10 | 5 | 3
Fatigue (General disorders) | 6 | 3 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 5 | 1 | 1 | 0
Pyrexia (General disorders) | 12 | 8 | 6 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 14 | 1 | 9 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 20 | 5 | 9 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 3 | 4 | 0
Bilirubin conjugated increased (Investigations) | 8 | 1 | 5 | 0
Blood bilirubin increased (Investigations) | 13 | 1 | 11 | 0
Blood phosphorus decreased (Investigations) | 1 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 8 | 0 | 3 | 0
Haemoglobin decreased (Investigations) | 3 | 8 | 3 | 0
Platelet count decreased (Investigations) | 2 | 3 | 4 | 1
Weight increased (Investigations) | 3 | 3 | 4 | 1
White blood cell count increased (Investigations) | 1 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 2 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 3 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 10 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 4 | 3 | 1
Headache (Nervous system disorders) | 14 | 6 | 8 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 22 | 4 | 9 | 1
Hypertension (Vascular disorders) | 5 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.